CLINICAL TRIAL: NCT04133337
Title: One-arm Exploratory Study on the Efficacy and Safety of Apatinib Combined With SHR-1210 Injection (PD-1 Antibody) in the Treatment of Removable IB-IIIA Non-small Cell Lung Cancer
Brief Title: Apatinib Combined With SHR-1210 Injection in the Treatment of Patients With Removable IB-IIIA NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Juan LI, MD, MD, Sichuan Cancer Hospital and Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-SHR-NSCLC201906
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Lung Diseases; Neoplasms; Respiratory Tract Diseases; Thoracic Neoplasms; Non-small-cell Lung Cancer
Keywords: Apatinib; SHR-1210; NSCLC; neoadjuvant
MeSH Terms: conditions — Lung Diseases; Neoplasms; Respiratory Tract Diseases; Thoracic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib Combined With SHR-1210 Injection (Experimental): * Drugs:Apatinib Apatinib mesylate tablets 250 mg qd po, discontinued one week before surgery.
  * Drugs: SHR-1210 SHR-1210 injection 200mg (5mL), ivgtt, q2w, 3 cycles, each time 20-60min completed infusion.
  * Surgery:
  The patient underwent imaging examinations within 7 days prior to surgery, including chest CT and related metastatic examinations. The patient underwent surgery 7-8 weeks after the first dose.
  Interventions: Drug: Apatinib; Drug: SHR-1210

INTERVENTIONS:
Drug: Apatinib — Apatinib Mesylate Tablets
  Other Names: AiTan; H20140103
Drug: SHR-1210 — Camrelizumab for Injection
  Other Names: Camrelizumab; Karuilizhu Dankang; S20190027

SUMMARY:
The aim of this study was to investigate the safety and efficacy of SHR-1210 in combination with the anti-vascular survival target drug apatinib in patients with resectable NSCLC, and to provide new treatment options for neoadjuvant therapy in patients with the period IB-IIIA NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 years old to 75 years old, male or female;
* 2. Initial treatment of patients with IB-IIIA non-small cell lung cancer who are expected to be surgically resected;
* 3. Histopathologically confirmed non-small cell lung cancer with measurable tumor lesions (spiral CT scan≥10mm, meeting RECIST 1.1 criteria);
* 4. ECOG PS: 0-1 points
* 5. The function of important organs meets the following requirements (no blood components and cell growth factors are allowed for 2 weeks before the start of study): Absolute neutrophil count (ANC)≥1.5×10 E+9/L; platelets≥100×10E+9/L / L; hemoglobin ≥9g/dL; serum albumin(ALB)≥2.8g/dL; a total bilirubin (TBil) of≤1.5 ULN, ALT and AST≤2.5 ULN, in case of liver metastasis, ALT and AST≤5 ULN; creatinine clearance rate≥ 50mL/min(Cockcroft-Gault);thyroid function is normal.
* 6. Estimated survival time≥3 months;
* 7. Female subjects with fertility should undergo a urine or serum pregnancy test within 72 hours prior to the first study drug administration and are shown to be negative ,and willing to be 3 months after the last dose of SHR-1210 injection during the trial period. The effective method was used for contraception (from the control group to 180 days after the last administration). For male subjects whose partners are women of childbearing age, effective methods should be used during the test period and within 3 months after the last administration of SHR-1210 injection (control group to 180 days after the last administration);
* 8. Patients were voluntarily enrolled in the study and signed an informed consent form (ICF) with good adherence and follow-up.

Exclusion Criteria:

* 1. The patient has any active autoimmune disease or a history of autoimmune disease;
* 2.The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppression purposes (dose>10 mg / day of prednisone or other therapeutic hormones);
* 3.Interstitial pneumonia ;
* 4.Severe allergic reactions to other monoclonal antibodies ;
* 5.Suffering from high blood pressure and not being well controlled by antihypertensive medication (systolic blood pressure≥140 mmHg or diastolic blood pressure≥90 mmHg) ;
* 6.Have clinical symptoms or disease that are not well controlled ;
* 7.Abnormal coagulation function (INR>2.0, PT>16s), bleeding tendency or receiving thrombolysis or anticoagulant therapy, allowing prophylactic use of low-dose aspirin, low molecular weight heparin;
* 8.There was significant coughing blood in the first 2 months before enrollment, or daily hemoptysis amounted to 2.5ml or more;
* 9.Significant clinically significant bleeding symptoms or a clear tendency to hemorrhage during the first 3 months of randomization;
* 10.Urinary routine suggests urinary protein≥ ++ and confirmed 24-hour urine protein> 1.0 g ;
* 11.The patient has active infection, unexplained fever within 3 days before administration, ≥38.5 °C, or baseline white blood cell count>15×109/L;
* 12.The patient has previously received other PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1;
* 13.Other patients considered by the treating physician not suitable for inclusion .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response rate(MPR)(<10% viable tumor cells) | At time of surgery
  To assess the major pathologic response rate (<10% viable tumor cells) in patients receiving Apatinib Combined With SHR-1210 Injection.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 2 years
  the proportion of patients with a best overall response of CR, PR or SD in the whole body, as assessed per RECIST 1.1 by the investigator.
Overall response rate (ORR) | up to 2 years
  the proportion of patients with a best overall confirmed response of CR or PR in the whole body as assessed per RECIST 1.1 by the investigator
Disease-free survival (DFS) | up to 2 years
  Defined as the time from date of surgery until recurrence of tumor or death from any cause

OTHER OUTCOMES:
Incidence of irAEs | up to 2 years
  Grade 3 or higher per Common Terminology Criteria for Adverse Events (CTCAE V5.0)
Incidence of SAEs | up to 2 years
  Grade 3 or higher per Common Terminology Criteria for Adverse Events (CTCAE V5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, MD, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No